CLINICAL TRIAL: NCT06483334
Title: A Phase 1/2 Randomized, Umbrella Study to Evaluate the Efficacy and Safety of MK-2870 Plus Enfortumab Vedotin (EV) With and Without Pembrolizumab, as Treatment for Participants With Advanced Urothelial Carcinoma (KEYMAKER-U04): Substudy 04C
Brief Title: A Study of Efficacy and Safety of Sacituzumab Tirumotecan (MK-2870) Plus Enfortumab Vedotin (EV) With and Without Pembrolizumab in Advanced Urothelial Carcinoma (MK-3475-04C/KEYMAKER-U04)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-04C; MK-3475-04C (Other: MSD); 2023-506387-14-00 (Registry Identifier: EU CT); U1111-1293-7631 (Registry Identifier: UTN)
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Urothelial Carcinoma; Locally Advanced Urothelial Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Transitional Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Part 1 is non-randomized open-label. Part 2 is randomized open-label (as of Amendment 5, Part 2 will not be conducted).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab tirumotecan plus EV (Experimental): Participants will receive sacituzumab tirumotecan as an intravenous (IV) infusion and EV as an IV infusion on Days 1 and 8 of every 3-week cycle until disease progression, intolerable toxicity, or investigator decision.
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Enfortumab Vedotin; Drug: Supportive care measures
- Sacituzumab tirumotecan plus EV and pembrolizumab (Experimental): Participants will receive sacituzumab tirumotecan as an IV infusion and EV as an IV infusion on Days 1 and 8 of every 3-week cycle until disease progression, intolerable toxicity, or investigator decision. Participants will also receive pembrolizumab 200 mg as an IV infusion on Day 1 of every 3-week cycle for up to ~2 years (35 cycles).
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Enfortumab Vedotin; Biological: Pembrolizumab; Drug: Supportive care measures

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — IV infusion at different dose levels
  Other Names: MK-2870; SKB264
Biological: Enfortumab Vedotin — IV infusion at different dose levels
  Other Names: PADCEV™
Biological: Pembrolizumab — 200 mg IV infusion
  Other Names: MK-3475; KEYTRUDA
  Arms: Sacituzumab tirumotecan plus EV and pembrolizumab
Drug: Supportive care measures — Participants are allowed to take supportive care measures at the discretion of the investigator. Prophylactic supportive care measures may include but are not limited to antiemetic agents, antidiarrheal agents, granulocyte and erythroid growth factors, and blood transfusions.

SUMMARY:
This study is a substudy being conducted under one pembrolizumab umbrella master study KEYMAKER-U04. The substudy will consist of 2 parts. Part 1 will evaluate the safety and preliminary efficacy of sacituzumab tirumotecan plus enfortumab vedotin (EV). Part 2 will be based on Part 1 results and will evaluate the efficacy, pharmacokinetics, and safety of sacituzumab tirumotecan plus EV in combination with pembrolizumab in participants with advanced urothelial carcinoma.

DETAILED DESCRIPTION:
The master study for this substudy is MK-3475-U04/KEYMAKER-U04. The master study will not be screening any participants and will not be registered.

As of Amendment 5, Part 2 will not be conducted. No participants will be enrolled in Part 2, and no data for Part 2 will be collected.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Must have histologically documented, locally advanced/metastatic urothelial carcinoma (la/mUC).
* Must provide an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion demonstrating UC, not previously irradiated, and adequate for biomarker evaluation. A newly obtained biopsy is strongly preferred, but not required if archival tissue is evaluable.
* Any AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Endocrine-related AEs adequately treated with hormone replacement are eligible.
* PART 1 ONLY: Participants must have received platinum-based chemotherapy for treatment of la/mUC.
* PART 1 ONLY: Participants must not have received >2 lines of therapy for la/mUC. Platinum-based chemotherapy followed by avelumab maintenance is considered 2 lines of therapy.
* PART 2 ONLY: Participants must not have received prior systemic therapy for la/mUC.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Has Grade ≥2 peripheral neuropathy.
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing.
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea).
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease and/or serious cardiovascular and cerebrovascular diseases within the 6 months preceding study intervention.
* Has active keratitis or corneal ulcerations. Superficial punctate keratitis is allowed if the disorder is being adequately treated in the opinion of the investigator.
* Has a history of uncontrolled diabetes.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention.
* PART 2 ONLY: Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of study intervention. Inhaled or topical steroids are permitted in the absence of active autoimmune disease. Physiologic replacement doses of corticosteroids are permitted for participants with adrenal insufficiency.
* PART 2 ONLY: Has an active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy.
* Is human immunodeficiency virus (HIV)-infected and has a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Has active Hepatitis B or Hepatitis C virus infection.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* PART 2 ONLY: History of allogeneic tissue/solid organ transplant.
* Has not adequately recovered from major surgery or has ongoing surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Percentage of Participants with Dose-limiting toxicities (DLT) | Up to 21 days
  A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE 5.0). The number of participants who experience a DLT in Part 1 will be reported.
Part 1: Percentage of Participants Who Experienced At Least One Adverse Event (AE) | Up to ~3 years
  An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of participants experiencing an AE in Part 1 will be reported.
Part 1: Percentage of Participants Who Discontinued Study Treatment Due to an AE | Up to ~2 years
  An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of participants who discontinue study treatment due to an AE in Part 1 will be reported.
Part 2: Percentage of Participants with DLT | Up to 21 days
  A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the NCI CTCAE 5.0. The number of participants who experience a DLT in Part 2 will be reported.
Part 2: Percentage of Participants Who Experienced At Least One AE | Up to ~3 years
  An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of participants experiencing an AE in Part 2 will be reported.
Part 2: Percentage of Participants Who Discontinued Study Treatment Due to an AE | Up to ~2 years
  An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of participants who discontinue study treatment due to an AE in Part 2 will be reported.
Part 2: Objective Response Rate (ORR) | Up to ~3 years
  ORR is defined as the percentage of participants who achieve a confirmed complete response (CR) (disappearance of all target lesions) or partial response (PR) (at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by investigator. ORR will be reported for participants in Part 2.

SECONDARY OUTCOMES:
Part 1: ORR | Up to ~3 years
  ORR is defined as the percentage of participants who achieve a confirmed CR or PR per RECIST 1.1 as assessed by investigator. ORR will be reported for participants in Part 1.
Part 2: Duration of Response (DOR) | Up to ~3 years
  For participants who demonstrate confirmed CR or PR per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by investigator will be presented.
Part 1: Maximum Serum Concentration (Cmax) of Sacituzumab Tirumotecan-Antibody-Drug Conjugate (ADC) | Days 1, 8, 15 of Cycle 1 (each cycle is 21 days), Day 1 of Cycle 2, Days 1 and 8 of Cycle 3, Day 1 of Cycles 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Cmax of sacituzumab tirumotecan-ADC in Part 1.
Part 1: Serum Trough Concentration (Ctrough) of Sacituzumab Tirumotecan-ADC | Days 1, 8, 15 of Cycle 1 (each cycle is 21 days), Day 1 of Cycle 2, Days 1 and 8 of Cycle 3, Day 1 of Cycles 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Ctrough of sacituzumab tirumotecan-ADC in Part 1.
Part 1: Cmax of Free Payload for Sacituzumab Tirumotecan | Days 1, 8, 15 of Cycle 1 (each cycle is 21 days), Day 1 of Cycle 2, Days 1 and 8 of Cycle 3, Day 1 of Cycles 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Cmax of free payload for sacituzumab tirumotecan in Part 1.
Part 1: Ctrough of Free Payload for Sacituzumab Tirumotecan | Days 1, 8, 15 of Cycle 1 (each cycle is 21 days), Day 1 of Cycle 2, Days 1 and 8 of Cycle 3, Day 1 of Cycles 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Ctrough of free payload for sacituzumab tirumotecan in Part 1.
Part 1: Cmax of Enfortumab Vedotin-ADC | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycle 2, Days 1 and 8 of Cycle 3, and Day 1 of Cycles 4 and 8
  Blood samples collected at designated time points will be used to determine the Cmax of enfortumab vedotin-ADC in Part 1.
Part 1: Ctrough of Enfortumab Vedotin-ADC | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycle 2, Days 1 and 8 of Cycle 3, and Day 1 of Cycles 4 and 8
  Blood samples collected at designated time points will be used to determine the Ctrough of enfortumab vedotin-ADC in Part 1.
Part 1: Cmax of Free Payload for Enfortumab Vedotin | Days 1, 8, 15 of Cycle 1 (each cycle is 21 days), Day 1 of Cycle 2, Days 1 and 8 of Cycle 3, and Day 1 of Cycles 4 and 8
  Blood samples collected at designated time points will be used to determine the Cmax of free payload for EV in Part 1.
Part 1: Ctrough of Free Payload for Enfortumab Vedotin | Days 1, 8, 15 of Cycle 1 (each cycle is 21 days), Day 1 of Cycle 2, Days 1 and 8 of Cycle 3, and Day 1 of Cycles 4 and 8
  Blood samples collected at designated time points will be used to determine the Ctrough of free payload for EV in Part 1.
Part 1: Incidence of Antidrug Antibodies (ADA) to Sacituzumab Tirumotecan | Day 1 of Cycles 1 (each cycle is 21 days), 2, 3, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated timepoints will be used to determine the ADA response to sacituzumab tirumotecan. The incidence of ADAs over time in Part 1 will be presented.
Part 1: Incidence of ADA to Enfortumab Vedotin | Day 1 of Cycles 1 (each cycle is 21 days), 2, 3, 4 and 8
  Blood samples collected at designated timepoints will be used to determine the ADA response to sacituzumab tirumotecan. The incidence of ADAs over time in Part 1 will be presented.
Part 2: Cmax of Sacituzumab Tirumotecan-ADC | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycles 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Cmax of sacituzumab tirumotecan-ADC in Part 2.
Part 2: Ctrough of Sacituzumab Tirumotecan-ADC | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycles 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Ctrough of sacituzumab tirumotecan-ADC in Part 2.
Part 2: Cmax of Free Payload for Sacituzumab Tirumotecan | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycles 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Cmax of free payload for sacituzumab tirumotecan in Part 2.
Part 2: Ctrough of Free Payload for Sacituzumab Tirumotecan | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycles 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Ctrough of free payload for sacituzumab tirumotecan in Part 2.
Part 2: Cmax of Enfortumab Vedotin-ADC | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycles 2, 4 and 8
  Blood samples collected at designated time points will be used to determine the Cmax of enfortumab vedotin-ADC in Part 2.
Part 2: Ctrough of Enfortumab Vedotin-ADC | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycles 2, 4 and 8
  Blood samples collected at designated time points will be used to determine the Ctrough of enfortumab vedotin-ADC in Part 2.
Part 2: Cmax of Free Payload for Enfortumab Vedotin | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycles 2, 4 and 8
  Blood samples collected at designated time points will be used to determine the Cmax of free payload for EV in Part 2.
Part 2: Ctrough of Free Payload for Enfortumab Vedotin | Days 1 and 8 of Cycle 1 (each cycle is 21 days), Day 1 of Cycles 2, 4 and 8
  Blood samples collected at designated time points will be used to determine the Ctrough of free payload for EV in Part 2.
Part 2: Cmax of Pembrolizumab-ADC | Days 1 of Cycles 1 (each cycle is 21 days), 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Cmax of pembrolizumab-ADC.
Part 2: Ctrough of Pembrolizumab-ADC | Days 1 of Cycles 1 (each cycle is 21 days), 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Ctrough of pembrolizumab-ADC.
Part 2: Cmax of Free Payload for Pembrolizumab | Days 1 of Cycles 1 (each cycle is 21 days), 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Cmax of free payload for pembrolizumab.
Part 2: Ctrough of Free Payload for Pembrolizumab | Days 1 of Cycles 1 (each cycle is 21 days), 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated time points will be used to determine the Ctrough of free payload for pembrolizumab.
Part 2: Incidence of ADA to Sacituzumab Tirumotecan | Day 1 of Cycles 1 (each cycle is 21 days), 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated timepoints will be used to determine the ADA response to sacituzumab tirumotecan. The incidence of ADAs over time in Part 2 will be presented.
Part 2: Incidence of ADA to Enfortumab Vedotin | Day 1 of Cycles 1 (each cycle is 21 days), 2, 4 and 8
  Blood samples collected at designated timepoints will be used to determine the ADA response to EV. The incidence of ADAs over time in Part 2 will be presented.
Part 2: Incidence of ADA to Pembrolizumab | Day 1 of Cycles 1 (each cycle is 21 days), 2, 4 and 8 and every 4 cycles thereafter up to Cycle 35, at end of treatment, and at 30 days post last dose
  Blood samples collected at designated timepoints will be used to determine the ADA response to pembrolizumab. The incidence of ADAs over time be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (25):
- United States (8):
  - University of California San Francisco HDFCCC ( Site 4044), San Francisco, California
  - University of Chicago Medical Center ( Site 4037), Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center ( Site 4011), Indianapolis, Indiana
  - Dana-Farber Cancer Institute ( Site 4047), Boston, Massachusetts
  - Siteman Cancer Center ( Site 4038), St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai ( Site 4018), New York, New York
  - Cleveland Clinic-Taussig Cancer Center ( Site 4036), Cleveland, Ohio
  - Huntsman Cancer Institute-HCI Clinical Trials Office ( Site 4041), Salt Lake City, Utah
- Canada (2):
  - The Ottawa Hospital - General Campus ( Site 4105), Ottawa, Ontario
  - Princess Margaret Cancer Centre ( Site 4106), Toronto, Ontario
- Centre Hospitalier Lyon Sud ( Site 4606), Pierre-Bénite, Auvergne-Rhône-Alpes, France
- Israel (3):
  - Rambam Health Care Campus ( Site 4501), Haifa
  - Rabin Medical Center-Oncology ( Site 4504), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 4503), Ramat Gan
- Italy (3):
  - Ospedale San Raffaele-Oncologia Medica ( Site 4403), Milan, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 4405), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 4406), Napoli
- Nederlands Kanker Instituut - Antoni van Leeuwenhoek - NKI-AVL ( Site 4302), Amsterdam, North Holland, Netherlands
- South Korea (3):
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 4903), Seoul
  - Asan Medical Center-Department of Oncology ( Site 4901), Seoul
  - Samsung Medical Center ( Site 4902), Seoul
- Spain (2):
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 4767), Barcelona
  - Hospital Clinico San Carlos ( Site 4765), Madrid
- National Cheng Kung University Hospital-Clinical Trial Center ( Site 4803), Tainan, Taiwan
- St Bartholomew s Hospital ( Site 4206), London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26212&tenant=MT_MSD_9011